CLINICAL TRIAL: NCT04861831
Title: Power Centering for Seniors: A Multimodal Intervention to Improve Mobility and Quality of Life in Older Adults
Brief Title: Power Centering for Seniors
Acronym: PCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Department of Geriatric Medicine FELIX PLATTER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BASEC ID 2018-00067
Record Dates: First submitted 2021-04-09; First posted 2021-04-27 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-07

CONDITIONS: Healthy Aging; Mobility Limitation; Walking, Difficulty
Keywords: Elderly; Walking speed; Gait; Falls; Quality of life; Independent living; Gait analysis; Physical functional performance; Montral Cognitive Assessment; Multimodal exercise; Exercise movement techniques; Muscle strength; Postural balance; Tai chi; Qi gong
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: This delayed intervention trial begins as a parallel group design with the Delayed Intervention (Dl) group serving as a control arm comparison for the Immediate Intervention (II) group. There is no control intervention. The ll and the Dl groups will be assessed pre-intervention. After the 12-week intervention for the II group, resp. the waiting period for the DI group, the lI group will undergo their post-intervention assessment. At that time, the Dl group will undergo their 2nd pre-intervention assessment to document any change in baseline measures that may have occurred. No significant changes are expected, so that at the end of the trial, data from the ll and the Dl groups can be pooled to provide results on the overall changes in outcome measures for all participants post- versus pre-intervention. After the 2nd pre-intervention assessment, the Dl group will have their intervention, post-intervention assessment, follow-up period and final assessment, as with the II group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate PCS Intervention (Experimental): After the pre-intervention clinical assessments, immediate (within one week) begin with the PCS exercise program (75-minute group class, twice weekly for 12 weeks; home practice of exercises recommended but not required). Post-intervention clinical assessments within one week after the last intervention class, followed by a 12-week follow-up period (continuation of exercise program at home recommended but not required). Final clinical assessments within one week after the 12-week follow-up period.
  Interventions: Other: Power Centering for Seniors intervention
- Delayed PCS Intervention (Experimental): During the 12 weeks that the Immediate Intervention (II) group participates in the PCS intervention, the Delayed Intervention (DI) group waits (there is no control intervention) and serves as a control arm comparison for the II group during this time. After the 12 weeks, the DI group will undergo a second pre-intervention assessment to document any change in baseline measures that may have occurred in those 12 weeks. No significant changes are expected. The DI group then begins the same exercise intervention (75-minute group class, twice weekly for 12 weeks; home practice of exercises recommended but not required) that the II group underwent, given by the same instructors. Post-intervention clinical assessments, 12-week follow-up period, and final clinical assessments after the follow-up period as described for the II group. After the trial, pooled data from both groups will provide results on the overall changes in outcome measures post- versus pre-intervention.
  Interventions: Other: Power Centering for Seniors intervention

INTERVENTIONS:
Other: Power Centering for Seniors intervention — Power Centering for Seniors is an innovative East-meets-West intervention (75-minute, twice weekly, supervised group classes over 12 weeks) that integrates Western best practice muscle strength and balance training components with Chinese Tai Chi/Qi Gong to improve mobility and quality of life in older, community-dwelling adults. Home practice is recommended (approximately 30 minutes three times per week on non-course days). The modularly designed course consists of four cycles with six themes repeated in each cycle. Course exercises increase in intensity throughout the twelve-week intervention period. Repetition of cycles and themes prepares participants for continuing their individualized version of the program after the group course intervention is complete. This should lead to long-term practice of the exercises learned in the intervention and to sustained positive effects of the training.

SUMMARY:
Walking difficulties, mobility decline and falls are prevalent among older adults. The incidence of each of these increases with age and the presence of each can negatively affect the quality of life in older adults. The purpose of this prospective clinical trial is to evaluate the efficacy of the Power Centering for Seniors multimodal, twice weekly, 12-week group intervention program to improve the mobility and quality of life in older, community-dwelling adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older
* Community-dwellers (i.e. not living in a skilled care or other institution)
* Able to walk at least 5 meters with or without a walking aid but without the assistance of another person
* Normal (habitual, self-paced) walking speed 80-100 cm/s
* Montreal Cognitive Assessment score 18 or more points
* lnformed Consent as documented by signature

Exclusion Criteria:

* Clinically significant neurologic or musculoskeletal diseases which severely affect walking, e.g. advanced Parkinson's disease or hemiplegia
* Other clinically significant non-stable medical or psychiatric conditions (e.g., renal failure, hepatic dysfunction, cardiovascular disease, advanced chronic pulmonary disease, psychosis, schizoaffective disorder, etc.) that, according to the study investigators, could endanger the participant and/or negatively affect study adherence
* Terminal illness
* Fracture (exception: teeth) in the previous 3 months
* Blindness
* lnability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous participation in the Power Centering for Seniors program
* Current participation in another (non-observational) clinical study

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Gait speed | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Change in the ratio of post- to pre-intervention normal (habitual, self-selcted) walking speed (cm/s) in the immediate intervention group compared to the ratio of post- to pre-waiting normal walking speed in the delayed intervention group.

SECONDARY OUTCOMES:
Cadence | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Cadence (number of steps per minute) quantified during gait analysis using the GAITRite electronic walkway system
Base of support | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Base of support (cm), the distance between heels, quantified during gait analysis using the GAITRite electronic walkway system.
Step width variability | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Step width variability (%) quantified during gait analysis using the GAITRite electronic walkway system. Variability calculated by the coefficient of varation=(standard deviation/mean)x100.
Single support time | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Single support time (s), an indirect measure of dynamic balance and gait certainty, quantified during gait analysis using the GAITRite electronic walkway system
Double support time | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Double support time (s), an indirect measure of dynamic balance and gait certainty, quantified during gait analysis using the GAITRite electronic walkway system
Stride time | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Stride time (s), also referred to as gait cycle time, quantified during gait analysis using the GAITRite electronic walkway system
Stride time variability | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Stride time variability (percent) quantified during gait analysis using the GAITRite electronic walkway system. Variability calculated by the coefficient of varation=(standard deviation/mean)x100.
Swing time | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Swing time (s), the time one leg is in the air during one gait cycle, quantified during gait analysis using the GAITRite electronic walkway system.
Swing time variability | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Swing time variability (percent) quantified during gait analysis using the GAITRite electronic walkway system. Variability calculated by the coefficient of varation=(standard deviation/mean)x100.
Timed Up and Go Test | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Standardized assessment of general mobility in older adults, time measured in seconds using a stopwatch
Timed Up and Go Test, imagined | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  After performing the Timed Up and Go Test, the participant remains seated and imagines performing the Timed Up and Go Test. Test time is measured in seconds using a stopwatch. Time for imagined test performance that is twice as fast or faster than real test performance time reflect possible cognitive difficulties as well as walking difficulties, particularly under dual or multi-task conditions.
Short Physical Performance Battery | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Standardized assessment of physical performance with measurements of muscle strength, balance and walking. Results range from 0 to 12 points, higher point score represents better physical performance.
Continuous Scale of Physical Functional Performance Test | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Strandardized assessment of physical functional performance of 10 tasks of daily living. Task results measured as time (s), weight (kg) and/or distance (cm or m, depending on task) are transformed by the assessment software into scaled scores ranging from 0 to 100 points, with higher point scores reflecting better performance and greater liklihood of independent living. Total score (0-100 points) and well as subscores (0-100 points) of five domains of physical functional perfomance are provided: upper body strength, upper body flexibility, lower body strength, balance and coordination, and endurance
Physical Activity Scale for the Elderly | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Standardized, self-report questionnaire to measure physical activity levels in older people as well as to assess the effectiveness of exercise interventions. From a list of 12 types of activities and referring to the previous week, participants report how many days per week and for how many hours per day they performed each activity. Scores are calculated by multiplying the weight (activity weights are provided in a table for PASE scoring) by the frequency values for each of 12 types of activities. Scores may range from zero to 400 or more. Higher scores reflect higher levels of physical activity.
Grip strength | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Grip strength, as a surrogate marker of overall muscle strength, measured using a Martin vigorimater (kPa)
5x Sit to Stand Test | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  General functional measure of lower body strength, measured in seconds using a stop watch, performed as part of the Short Physical Performance Battery.
Modified Clinical Test of Sensory lnteraction and Balance | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Assesses balance under four test conditions. Time to perform each task is measured in seconds with a stopwatch, results range from not being able to perform a task to maximal task time of 30 seconds. Postural sway will be measured during each task with the APDM system (measured in angle, m/s2, Hz or m2/s4, depending on paramter)
Falls | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), and monthly throughout the trial duration for II and DI
  Fall incidence will be documented from the pre-intervention assessment until the end of the follow-up period via monthly diaries completed by study participants as well as via monthly phone calls with the study team.
Fear of falling | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Self-reported using the Falls Efficacy Scale-lnternational version (FES-I) questionnaire (scores range from 1 to 64 points, higher point scores reflect greater subjective fear of falling), as well as binary responses (yes/no) of participants at each clinical visit
Montreal Cognitive Assessment test | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  Standardized test of general cognition, administered by trained site staff. Scores range from 0 to 30 points, higher point scores reflect better cognition
Short Form-36, version 2, acute recall assessment of health-related quality of life | II Group: pre-intervention (Week 1), post-intervention (Week 12), post-follow-up (Week 24); DI Group: first pre-intervention (Week 1), second pre-intervention (Week 12), post-intervention (Week 24), post-follow-up (Week 36)
  This self-report questionnaire is a reliable and valid tool for measuring health-related quality of life. It consists of 36 questions (acute recall = previous week) reflecting eight domains of health and provides eight scaled scores, which are the weighted sums of the questions in each respective domain. Each scale is directly transformed into a score of 0 to 100 points on the assumption that each question carries equal weight. Lower scores are associated with greater disability and lower quality of life.
lntervention course attendance | At each course lesson (twice weekly throughout the 12 week intervention period) for the II and the DI group
  Number of intervention courses from maximum 24 that each participant attends, as a marker of intervention adherence, will be documented by course instructors at each class

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A. Bridenbaugh, M.D., Principal Investigator — University Department of Geriatric Medicine FELIX PLATTER
Locations (1):
- University Department of Geriatric Medicine FELIX PLATTER, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rossler R, Birrer M, Haslbauer A, Goldfarb J, De Spiegeleer A, Hardi I, Kressig RW. Efficacy of the power centering for seniors intervention on physical functional performance in older community-dwelling adults: a secondary analysis of a randomised controlled trial. Sci Rep. 2025 Aug 7;15(1):28908. doi: 10.1038/s41598-025-13404-6. PMID 40775497
- See also: study site website and trial description (in German) — https://www.felixplatter.ch/index
- See also: Power Centering for Seniors website of the Legacy of Wisdom Swiss Association — https://www.centeringforseniors.org/the-research-summary